CLINICAL TRIAL: NCT05307588
Title: Satisfaction With Life and Psychological Distress During the COVID-19 Pandemic: An Egyptian Online Cross-sectional Study
Brief Title: Psychological Distress During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Loutfy, Lecturer of Pediatric Nursing, Beni-Suef University
Other Study IDs: COVID-19
Record Dates: First submitted 2022-03-31; First posted 2022-04-01 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Psychological Distress; COVID-19 Pandemic; Satisfaction
Keywords: psychosocial effects; COVID-19
MeSH Terms: conditions — COVID-19; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Design, sample, and setting This is a cross-sectional study using an Internet-based self-administered questionnaire of closed-ended questions and using convenience sampling. In total, 612 undergraduate students completed the survey in Mansoura University.

Data collection Data was collected anonymously through an online questionnaire created using the technology of Google Forms provided by Google ™ and was constructed in Arabic language. The questionnaire consisted of three sections. The first section assessed students' baseline characteristics including sex, age, area of study, academic level, residence, marital status, family members infected, close people infected, and knowing someone who died of the infection.

The second section measured the psychosocial effects of COVID-19 pandemic using two instruments, University of California Los Angeles (UCLA) Loneliness Scale, version 324 and Depression Anxiety Stress Scale (DASS-21).19 The UCLA Loneliness Scale is a widely used self-report instrument of loneliness consisting of 20 items designed to measure both emotional as well as social loneliness. Response of each item was rated on a four-point scale from (1) never to (4) always felt as expressed in each item. Final score ranges from 20 to 80 with higher scores demonstrating higher feelings of loneliness. The scale's reliability was found to be high with alpha coefficients ranging from 0.89 to 0.94 for samples of students. The Arabic version of UCLA Loneliness Scale was used in the current study according to the Arabic translation in Egyptian culture by Daswqee.20 The correlation coefficients values were 0.76 for females and 0.74 for males.

DETAILED DESCRIPTION:
Since December 2019, the novel coronavirus disease 2019 (COVID-19) has spread from Wuhan city to different areas in China and around the world. On 11 March 2020, the World Health Organization (WHO) declared the COVID-19 outbreak a pandemic. On 14 February 2020, the Egyptian Ministry of Health reported the first case of COVID-19. To control the COVID-19 outbreak, the Egyptian government introduced preventive and containment measures with a partial closure starting on 25 March. On 31 March, Egypt pronounced 710 COVID-19 cases and 46 related deaths with a mortality rate of 6.48%. As on 06 June 2020, there were 1497 new cases with total cases of 32 612, a total of 1198 deaths and 8538 full recovery. Generally, several potential stressors were caused by the pandemic that might lead to psychological distress and life dissatisfaction. Individuals' overall assessments of their psychological wellbeing and quality of life are referred to as life satisfaction. Psychological distress takes the shape of a negative emotion, which contrasts with life contentment. It refers to people's unfavorable emotional reactions to several stimuli, which might include tension, dread, worry and psychological instability.

ELIGIBILITY:
Inclusion Criteria:

- All available adults can fill in online surveys.

Exclusion Criteria:

- Children under 18 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - adults (18 years and above) in all regions of Egypt who were willing to participate in the study. The study adopted an online survey, and the study population may not reflect the actual pattern of the general population.
Sampling Method: Non-Probability Sample
Enrollment: 1056 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Measuring the levels of psychological distress. | Within one week (06 to 13 June 2020).
  A 10-item 5-point scale (10-50 score) is a self-report questionnaire used for measuring the levels of psychological distress. The respondents choose the most relevant response for them in the last 4 weeks. After summing scores, the range of 10-15, 16-21, 22-29 and 30-50 represent low, moderate, high and very high psychological distress, respectively
Satisfaction with Life Scale | Within one week (06 to 13 June 2020).
  A self-report questionnaire intended to determine the level of satisfaction with life composed of 5-item rated on 7-point scale. After summing scores, the range of 5-9, 10-14, 15-19, 21-25, 26-30 and above 31 reflect extremely dissatisfied, dissatisfied, slightly dissatisfied, slightly satisfied, satisfied, and extremely satisfied with life, respectively. A score of 20 reflects the impartial point on the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Loutfy, PhD, Principal Investigator — Department of Pediatric Nursing, Faculty of Nursing- Beni Suef University, Egypt; Moustafa Saad, PhD, Principal Investigator — Department of Gerontological Nursing, Faculty of Nursing-Mansoura University, Egypt; Ahmed Ali, PhD, Principal Investigator — Department of Pediatric Nursing, Faculty of Nursing- Mansoura University, Egypt; Abdel-Hady El-Gilany, PhD, Principal Investigator — Department of Public Health and Preventive Medicine, Faculty of Medicine, Mansoura University, Egypt; Mohamed Zoromba, PhD, Principal Investigator — Department of Psychiatric and Mental Health Nursing, Faculty of Nursing-Mansoura University, Egypt
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, Ho RC. Immediate Psychological Responses and Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19) Epidemic among the General Population in China. Int J Environ Res Public Health. 2020 Mar 6;17(5):1729. doi: 10.3390/ijerph17051729. PMID 32155789